CLINICAL TRIAL: NCT05276310
Title: An Open-Label, Dose-Escalation and Expansion, Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of IMC-002 in Patients With Advanced Cancer Failed to Standard Therapy
Brief Title: A Study of IMC-002 in Patients With Advanced Cancer Failed to Standard Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneOncia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMC-002-K102
Record Dates: First submitted 2022-02-22; First posted 2022-03-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Advanced Cancer
Keywords: IMC-002; Phase I; CD47; SIRPα

STUDY DESIGN:
Intervention Model Description: Part 1: Dose Escalation Part 2: Expansion cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMC-002 (Experimental): IMC-002
  Interventions: Biological: IMC-002

INTERVENTIONS:
Biological: IMC-002 — Part 1: Dose escalation IMC-002 5, 10, 20, and 30 mg/kg over 3 hours (±30 minutes) intravenous (IV) infusion every 2 weeks Part 2: Expansion cohort IMC-002 20 mg/kg over 3 hours (±30 minutes) IV infusion at the first cycle, if the first infusion is tolerated, then over 1 to 1.5 hours (±10 minutes) IV infusion at all following cycles every 3 weeks In hepatocellular (HCC) Cohort, Lenvatinib 8 mg once daily (body weight of < 60 kg), or 12 mg once daily (body weight of ≥ 60 kg) In triple negative breast cancer (TNBC) Cohort, Paclitaxel 175 mg/m2 IV infusion on Day 1 of each cycle, or Gemcitabine 1,000 mg/m2 followed by Carboplatin AUC 2 IV infusion on Day 1 and Day 8 of each cycle In biliary tract cancer (BTC) Cohort, Lenvatinib 8 mg once daily (body weight of < 60 kg), or 12 mg once daily (body weight of ≥ 60 kg) In B-cell lymphoma Cohort, Rituximab 375 mg/m2 IV infusion on Day 1 of each cycle

SUMMARY:
This is an Open-Label, Dose-Escalation and Expansion, Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of IMC-002 in Patients with Advanced Cancer Failed to Standard Therapy

DETAILED DESCRIPTION:
The purpose of this study is to evaluate safety and tolerability and to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of IMC-002.

Multiple-dose levels of IMC-002 will be tested in subjects with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. Adult (19 years or older)
3. Diagnosis and prior therapies

   3-1. Part 1: Histologically or cytologically proven metastatic or locally advanced solid tumors

   3-2. Part 2, HCC Cohort:
   1. Histologically or cytologically proven metastatic or locally advanced of hepatocellular carcinoma (excluding fibrolamellar, sarcomatoid or mixed cholangio-HCC tumors)
   2. Received ≥1 prior systemic therapy; lenvatinib-naive and eligible for lenvatinib.
   3. Child Pugh classification A

   3-3. Part 2, TNBC Cohort:
   1. Histologically or cytologically proven metastatic or locally advanced of triple negative breast cancer: negative of estrogen receptor (ER), progesterone receptor (PgR), and human epidermal growth factor receptor 2 (HER2)
   2. Received ≥1 prior systemic regimen and eligible for paclitaxel or gemcitabine/carboplatin. Patients who have previously received the planned SOC in this study (paclitaxel or gemcitabine/carboplatin) cannot be enrolled. If at least 6 months have elapsed since the completion of a prior SOC (paclitaxel, gemcitabine, and/or carboplatin) and the patient showed a tumor response to that regimen, the same SOC can be used in this trial.
   3. Bisphosphonate or denosumab for bone metastases is allowed if started before Cycle 1 Day 1. Prophylactic use of bisphosphonates or denosumab in patients without bone diseases is not permitted, except for the treatment of osteoporosis.

   3-4. Part 2, BTC Cohort:
   1. Histologically or cytologically proven metastatic or locally advanced of biliary tract cancer (gallbladder cancer, cholangiocarcinoma)
   2. Received ≥1 prior systemic therapy; lenvatinib-naive and eligible for lenvatinib

   3-5. Part 2, B-cell lymphoma Cohort:
   1. Histologically or cytologically proven CD20+ mature B-cell lymphoma according to 2016 WHO classification including:

      * diffuse large B-cell lymphoma (de novo or transformed)
      * Mantle cell lymphoma
      * Follicular lymphoma
      * Marginal zone lymphoma (nodal, extranodal or mucosa associated)
   2. Received ≥2 prior systemic therapies and eligible for rituximab treatment

      * For all cancer type, neo-adjuvant and/or adjuvant chemotherapy is not regarded as chemotherapeutic regimen for metastatic or recurrent cancer unless recurrence within 6 months after the last dose of anti-cancer drugs as neo-adjuvant and/or adjuvant therapy.
4. Subject must have at least 1 measurable lesion by RECIST 1.1
5. Availability of tumor archival material or fresh biopsies
6. ECOG performance status 0 or 1 and life expectancy ≥3 months
7. Adequate hematologic function, hepatic function, and renal function
8. Prior RT permitted if measurable disease exists outside the RT field or if disease progressed post-RT. RT must be completed ≥4 weeks before Cycle 1 Day 1
9. Agree to use effective contraception
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Treatment with nonpermitted drugs
2. Prior treatment with a CD47 or SIRPα targeting agent
3. Concurrent anticancer treatments
4. Major surgery or significant traumatic injury prior to Screening or planned major surgery during the study period
5. Previous malignant disease other than the target malignancy for this study
6. Active infection requiring systemic therapy before Day 1
7. Any active autoimmune disease, or history of autoimmune disease
8. Any psychiatric or cognitive condition
9. Known severe hypersensitivity reaction
10. Pregnant or lactating
11. Currently enrolled in another clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | 21 days
  To determine maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of IMC-002
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  * clinically significant changes in physical examination, vital signs, ECG parameters, clinical laboratory tests, AEs
  * Immunogenicity: anti-IMC-002 antibody

SECONDARY OUTCOMES:
Pharmacokinetics Endpoint : Cmax | through study completion, an average of 1 year
  maximum observed serum concentration (Cmax) of IMC-002
Pharmacokinetics Endpoint : Ctrough | through study completion, an average of 1 year
  minimum observed serum concentration immediately before dosing (Ctrough) of IMC-002
Pharmacokinetics Endpoint : Tmax | through study completion, an average of 1 year
  time of the maximum observed serum concentration (Tmax) of IMC-002
Pharmacokinetics Endpoint : AUC | through study completion, an average of 1 year
  Area Under the Serum Concentration-Time Curve (AUC) of IMC-002
Pharmacokinetics Endpoint : CL | through study completion, an average of 1 year
  total body clearance (CL) of IMC-002
Pharmacokinetics Endpoint : t½ | through study completion, an average of 1 year
  terminal half-life (t½) of IMC-002
Efficacy endpoints based on tumor assessment (Part2) : BOR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  best overall response (BOR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by RECIST 1.1 (for solid tumors) or Lugano criteria (for B-cell lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : ORR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  objective response rate (ORR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by RECIST 1.1 (for solid tumors) or Lugano criteria (for B-cell lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : DCR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  disease control rate (DCR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by RECIST 1.1 (for solid tumors) or Lugano criteria (for B-cell lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : DOR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  duration of response (DOR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by RECIST 1.1 (for solid tumors) or Lugano criteria (for B-cell lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : TTP | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  time-to-progression (TTP) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by RECIST 1.1 (for solid tumors) or Lugano criteria (for B-cell lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : PFS | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  progression-free survival (PFS) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by RECIST 1.1 (for solid tumors) or Lugano criteria (for B-cell lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : iBOR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  Immune best overall response(iBOR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by iRECIST(Solid tumor) or Lugano criteria with LYRIC modification(B-cell Lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : iORR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  Immune objective response rate(iORR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by iRECIST(Solid tumor) or Lugano criteria with LYRIC modification(B-cell Lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : iDCR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  Immune disease control rate(iDCR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by iRECIST(Solid tumor) or Lugano criteria with LYRIC modification(B-cell Lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : iDOR | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  Immune duration of response(iDOR) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by iRECIST(Solid tumor) or Lugano criteria with LYRIC modification(B-cell Lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : iTTP | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  Immune time-to-progression(iTTP) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by iRECIST(Solid tumor) or Lugano criteria with LYRIC modification(B-cell Lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : iPFS | Tumor assessments will be conducted every 2 cycles by contrast-enhanced CT (solid tumor), and every 3 cycles by PET-CT/CT with contrast (B-cell lymphoma), within 5 days prior to Day 1 of the next cycle, through study completion, an average of 1 year.
  Immune progression-free survival(iPFS) To evaluate efficacy of IMC-002 in combination with standard of care (SOC) anti-cancer therapy, as assessed by iRECIST(Solid tumor) or Lugano criteria with LYRIC modification(B-cell Lymphoma).
Efficacy endpoints based on tumor assessment (Part2) : overall survival (OS) | through study completion, an average of 1 year
  overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: HEUNG TAE KIM, MD, Study Director — ImmuneOncia Therapeutics Inc.
Locations (3):
- South Korea (3):
  - National Cancer Center, Ilsan
  - Asan Medical Center, Republic of Korea, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No